CLINICAL TRIAL: NCT06274398
Title: A Double-Blind, Placebo-Controlled, Randomized Phase 1 Study to Evaluate the Safety and Pharmacokinetics of Rectally Administered Tenofovir Alafenamide/Elvitegravir Inserts
Brief Title: Rectal Insert TAF/EVG Pre-Exposure Prophylaxis (RITE PrEP) Study
Acronym: RITE PrEP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: CONRAD (Other); Emory University (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: RITE Study
Record Dates: First submitted 2024-01-31; First posted 2024-02-23 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-02

CONDITIONS: Safety Issues
Keywords: rectal insert; HIV; pre-exposure prophylaxis (PrEP)

STUDY DESIGN:
Intervention Model Description: Randomized, Placebo-controlled, Double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): 2 TAF/EVG (20/16mg) rectal inserts
  Interventions: Drug: TAF/EVG rectal insert
- Placebo (Placebo Comparator): 2 Matching placebo inserts
  Interventions: Drug: Matching placebo rectal insert

INTERVENTIONS:
Drug: TAF/EVG rectal insert — Phase 1: rectal inserts applied daily for 3 consecutive days Phase 2: rectal inserts applied every other day for 14 days
  Arms: Active
Drug: Matching placebo rectal insert — Phase 1: rectal inserts applied daily for 3 consecutive days Phase 2: rectal inserts applied every other day for 14 days
  Arms: Placebo

SUMMARY:
This is a double-blind, placebo-controlled, randomized two-phase study to evaluate the safety and pharmacokinetics (PK) of two TAF/EVG inserts administered rectally for 3 consecutive days, then every other day for 14 days.

DETAILED DESCRIPTION:
The purpose of this study is to collect data regarding the safety and pharmacokinetics of repeat dosing schedules of TAF and EVG administered rectally to inform the development of future studies to assess the efficacy of this drug combination and mode of administration for use as on-demand PrEP in individuals at risk of acquiring HIV-1 infection.

Eligible participants will be stratified according to sex assigned at birth and then randomized 1:1 to either receive TAF/EVG inserts or placebo for self-administration during the study phases. During Phase 1, participants will self-administer two TAF/EVG or placebo rectal inserts for 3 consecutive days and return to the clinic at 24, 48, and 72 hours after the last dose for biological sample collection. During Phase 2, participants will administer two TAF/EVG or placebo rectal inserts every other day for 7 doses and return to the clinic at 24 hours, 48 hours, 72 hours and 7 days after the final dose for biological sample collection. There will be a washout period of 7 to 28 days between the study phases.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals between the ages of 18-59 years
2. Able to understand and give informed consent
3. HIV-negative and willing to be tested for HIV
4. Willing to undergo peripheral blood, urine, rectal secretion collection, and rectal biopsy sampling
5. For those assigned female at birth: Willing to undergo cervicovaginal secretion collection
6. Lifetime history of receptive anal intercourse
7. No contraindication to rectal biopsy (at the investigator's discretion)
8. For participants of childbearing potential: Willing to use an effective method of contraception for at least 30 days prior to enrollment and for the duration of study participation. Effective methods include:

   1. Hormonal methods
   2. Intrauterine device (IUD) inserted at least 30 days prior to enrollment
   3. Sterilization (of participant or partner)
   4. Sexually abstinent as defined by abstaining from penile-vaginal intercourse for 90 days prior to enrollment and intending to remain abstinent for the duration of study participation
   5. Willing to commit to using condoms for the duration of the study

Exclusion Criteria:

1. Currently infected with hepatitis virus and/or has liver disease
2. Current or chronic history of kidney disease or CrCl <60 ml/min
3. History of inflammatory bowel disease or other inflammatory, infiltrative, infectious, or vascular condition of the lower GI tract which at the judgement of the investigator, may be worsened by study procedures or may significantly distort the anatomy of the distal large bowel.
4. Significant laboratory abnormalities at baseline, including but not limited to:

   1. Hemoglobin ≤ 10 g/dL
   2. Platelet count <100,000
   3. Aspartate aminotransferase (AST) or alanine transaminase (ALT) >1.3x ULN
   4. Serum creatinine >1.3x upper limit of normal (ULN)
   5. PTT > 1.5x ULN or International normalized ratio (INR) >1.5x ULN
5. Any known medical condition that, in the judgement of the investigators, increases the risk of local or systemic complications of biopsy procedures or pelvic examination, including but not limited to:

   1. Uncontrolled or severe cardiac arrhythmia
   2. Recent major abdominal, cardiothoracic, or neurological surgery in the last 12 months
   3. History of uncontrolled bleeding diathesis
6. Current colonic, rectal, or cervicovaginal perforation, fistula, or malignancy
7. Current symptoms or evidence on clinical examination of ulcerative, suppurative, or proliferative lesions of the cervicovaginal and/or anorectal mucosa
8. Current symptoms or evidence on clinical examination of atypical rectal or vaginal discharge
9. Continued need for, or use during the 14 days prior to the rectal biopsy, of the following medications:

   1. Aspirin or more than 4 doses of NSAIDs
   2. Warfarin, heparin (LMW or unfractionated), platelet aggregation inhibitors, or fibrinolytic agents
   3. Any form of rectally administered medications or agents (excluding lubricants or douching)
10. Continued need for, or use during the 90 days prior to enrollment, of the following medications:

    1. Systemic immunomodulatory agents
    2. Supraphysiologic doses of steroids, except for short course steroids <7 days duration, at the discretion of the investigator
    3. Experimental medications, vaccines, or biologicals (except for COVID-19 vaccines available through the emergency use authorization)
11. Use of moderate or strong CYP inducers/inhibitors (see appendix I)
12. Known or suspected allergy to study product components
13. Use of pre-exposure prophylaxis (PrEP) for HIV prevention within 3 months prior to enrollment, and/or anticipated use and/or unwillingness to abstain from PrEP during trial participation
14. Use of post-exposure prophylaxis (PEP) for potential HIV exposure within 6 months prior to enrollment
15. Pregnant and breastfeeding persons, or intent to become pregnant within the next 6 months
16. Participation in other studies involving the use of drugs, medical devices, rectal and genital products, or vaccines within the past 90 days.
17. Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the participant unsuitable for the study or unable to comply with the study requirements.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Frequency and intensity of Adverse Events | from enrollment until Day 57 (after last rectal dose administration of study product)
  Safety measured by Grade 2 and higher adverse events (AEs)
Pharmacokinetics (PK) (maximum concentration (Cmax)) in blood | baseline and at 24, 48, and 72 hours after last rectal dose administration of study product in each Dosing Phase.
  concentrations of TFV-DP and EVG
PK (Cmax) in rectal secretions | baseline and at 24, 48, and 72 hours after last rectal dose administration of study product in each Dosing Phase.
  concentrations of TFV-DP and EVG
PK (Cmax) in rectal mucosal tissue | at 24 and 72 hours after last rectal dose administration of study product in each Dosing Phase.
  concentrations of TFV-DP and EVG

SECONDARY OUTCOMES:
PK (Cmax) in cervicovaginal secretions | at baseline and at 24, 48, and 72 hours after last rectal dose administration of study product in each Dosing Phase.
  concentrations of TFV and EVG
PK (Cmax) in cerviocovaginal mucosal tissues | at 24 hours after last rectal dose administration of study product in each Dosing Phase.
  concentrations TFV-DP and EVG
Cytokine Profiles | at baseline and at 24, 48, and 72 hours after last rectal dose administration of study product in Dosing Phases 1 and 2
  To assess a change in cytokine profiles in rectal and vaginal secretions
Microbiome Profiles | at baseline and at 24, 48, and 72 hours after last rectal dose administration of study product in Dosing Phases 1 and 2
  To assess a change to the microbiome composition in rectum and vagina

CONTACTS AND LOCATIONS:
Overall Officials: Cassie Grimsley Ackerley, MD, MSc, Principal Investigator — Emory School of Medicine; Richard E Haaland, Study Chair — Centers for Disease Control and Prevention; Gustavo F Doncel, MD, PhD, Study Chair — CONRAD
Locations (1):
- Emory Clinic, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No